CLINICAL TRIAL: NCT06190249
Title: A Phase I Study to Assess the Efficacy and Safety of Autologous Tumor Infiltrating Lymphocytes (LN144) With Adjuvant Pembrolizumab for Treatment of Immunotherapy Naïve Patients With High Risk Stage IIIb-dResectable Melanoma
Brief Title: Efficacy & Safety for LN144 With Pembrolizumab With High Risk Stage IIIb-dResectable Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Iovance withdrew support due to length of time required to meet accrual goal.
Sponsor: James Isaacs, MD (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, James Isaacs, MD, MD, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4622
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IIID Melanoma
Keywords: Autologous Tumor Infiltrating Lymphocytes; LN144; Resectable Melanoma; Immunotherapy Naive
MeSH Terms: conditions — Melanoma | interventions — lifileucel; Cyclophosphamide; Mesna; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LN-144 Therapy (Experimental): All patients will receive LN-144 therapy, consisting of these steps:
  1. Harvest (surgical resection of tumor tissue) to provide the autologous tissue that serves as the source of LN-144.
  2. Production of LN-144 investigational product (IP) at a central Good Manufacturing Practice (GMP) facility
  3. A 5-day nonmyeloablative lymphodepletion (NMA-LD) preparative regimen
  4. Infusion of the LN-144 product (Day 0)
  5. Administration of IV interleukin-2 (IL-2) for ≤ 6 doses.
  6. Infusion of pembrolizumab 200 mg (Week 12) every 3 weeks for up to 1 year (17 cycles)
  Interventions: Biological: LN-144; Drug: Cyclophosphamide; Drug: Mesna; Drug: Fludarabine; Biological: Interleukin-2 (IL-2); Drug: Pembrolizumab

INTERVENTIONS:
Biological: LN-144 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepleting chemotherapy including cyclophosphamide and fludarabine, patient is infused with autologous TIL (LN-144), followed by IL-2.
  Other Names: Autologous Tumor Infiltrating Lymphocytes (TIL)
Drug: Cyclophosphamide — Given by IV.
  Other Names: Cytoxan
Drug: Mesna — Given by IV.
  Other Names: Mesnex
Drug: Fludarabine — Given by IV.
  Other Names: Fludara
Biological: Interleukin-2 (IL-2) — Given by IV.
  Other Names: Aldesleukin; Proleukin
Drug: Pembrolizumab — Given by IV.
  Other Names: Keytruda

SUMMARY:
The purpose of this study is to evaluate the efficacy of adjuvant adoptive cell therapy (ACT) via infusion of LN-144 (autologous TIL) followed by interleukin-2 (IL-2) after a nonmyeloablative lymphodepletion (NMA-LD) preparative regimen, followed by Pembrolizumab.

DETAILED DESCRIPTION:
Primary:

• To evaluate the efficacy of LN-144 with adjuvant Pembrolizumab in Stage IIIb-d melanoma patients as assessed by 6 and 12-month relapse-free survival (RFS)

Secondary:

* To further evaluate the efficacy of LN-144 with adjuvant Pembrolizumab in Stage IIIb-d melanoma patients using overall survival (OS) and distant metastasis-free survival
* To characterize the safety profile of LN-144 in Stage IIIb-d melanoma patients as measured by the incidence of Grade ≥ 3 treatment emergent adverse events (TEAEs) within 3 months of LN-144 administration
* To identify location of relapse
* Rate of achievable recruitment for duration of planned recruitment period

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of resectable, Stage III, High-Risk melanoma defined by AJCC v8 as Stage IIIB, IIIC, or IIID.
* Disease must be resected to no evidence of disease on imaging and no gross disease residually with the exception of positive microscopic margin. No prior treatment with immunotherapy.
* One (1) lesion at least 1.5cm in size (solitary or aggregate) available for TIL harvesting that has not undergone prior embolization or RT in prior 3 months unless subsequent growth is demonstrated.
* Palliative radiation therapy is permitted so long as it does not involve lesions being selected for TIL. Washout is not required if all related toxicities have resolved to ≤ Grade 1 as per CTCAE v 5.0
* Previous surgical procedure(s) is/are permitted provided that wound healing has occurred, all complications have resolved, and at least 14 days have elapsed (for major operative procedures) prior to the tumor resection.
* Patients must have a washout period ≥ 21 days from prior anti-cancer therapy(ies) to the start of the planned NMA-LD pre-conditioning regimen.
* Patients must be ≥ 18 years of age at the time of consent.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and an estimated life expectancy of ≥ 3 months in the opinion of the Investigator.
* Patients must have the following hematologic parameters:• Absolute neutrophil count (ANC) ≥ 1000/mm3, •Hemoglobin (Hb) ≥ 9.0 g/dL, •Platelet ≥ 100,000/mm3
* Patients must have adequate organ function: •Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (≤ 3 × ULN); patients with liver metastasis ≤ 5 × ULN, •Estimated creatinine clearance (eCrCl) ≥ 40 mL/min using the Cockcroft-Gault formula at Screening, •Total bilirubin ≤ 2 mg/dL, •Patients with Gilbert's syndrome must have a total bilirubin ≤ 3 mg/dL
* Patients of childbearing potential (or female partners of male participants) must be willing to take the appropriate precaution to avoid pregnancy or fathering a child for the duration of the study and practice an approved, highly effective method of birth control during treatment and for 12 months after their last dose of IL-2.
* Approved methods of birth control are as follows: Combined (estrogen and progesterone containing) hormonal birth control associated with inhibition of ovulation: oral, intravaginal, transdermal, Progesterone-only hormonal birth control associated with inhibition of ovulation: oral, injectable, implantable, Intrauterine device (IUD), Intrauterine hormone-releasing system (IUS), Bilateral tubal occlusion, Vasectomized partner, True sexual abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar ovulation, symptothermal, post-ovulation methods) is not acceptable
* Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an ICF approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), and agree to abide by the study restrictions and return to the site for the required assessments, including the OS Follow-up Period.

Exclusion Criteria:

* Patients who have received an organ allograft or prior cell transfer therapy within the past 20 years that included a non-myeloablative or myeloablative chemotherapy regimen.
* Patients with melanoma of uveal/ocular origin.
* Patients who have a history of hypersensitivity to any component or excipient of LN-144 or other study drugs:

  * NMA-LD preparative regimen (cyclophosphamide, mesna, and fludarabine),
  * Proleukin®, aldesleukin, IL-2,
  * Pembrolizumab,
  * Antibiotics (ABX) of the aminoglycoside group (i.e., streptomycin, gentamicin); except those who are skin-test negative for gentamicin hypersensitivity,
  * Any component of the LN-144 infusion product formulation including dimethyl sulfoxide (DMSO), human serum albumin (HSA), IL-2, and dextran-40.
* Patients with symptomatic and/or untreated brain metastases (of any size and any number).
* Patients who are on chronic systemic steroid therapy except for those requiring steroid therapy for management of adrenal insufficiency; these patients may receive no more than 10 mg of prednisone or its equivalent daily.
* Patients who are pregnant or breastfeeding.
* Patients who have active medical illness(es) that would pose increased risk for study participation, including: active systemic infections requiring systemic ABX, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory, or immune systems.
* Patients must have a negative syphilis assay (per local standard, e.g., rapid plasma reagin [RPR], venereal disease research laboratory [VDRL]) and be seronegative for the human immunodeficiency virus (HIV1 and HIV2 antibody titers). Patients with positive serology for hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (anti-HBc) or hepatitis C virus (anti-HCV) indicating acute or chronic infection must have the corresponding polymerase chain reaction (PCR) assay; patients may be enrolled if the viral load by PCR is undetectable with/without active treatment. Additional serology testing may be required depending on local prevalence of certain viral exposures
* Patients who have any form of primary immunodeficiency (e.g., severe combined immunodeficiency disease [SCID] and acquired immunodeficiency syndrome [AIDS])
* Patients who have received a live or attenuated vaccination within 28 days prior to the start of NMA-LD pre-conditioning regimen.
* Participant has an LVEF < 45% and is New York Heart Association (NYHA) Class 1. For participants ≥ 60 years of age OR who have a history of clinically relevant cardiac disease, no irreversible wall movement abnormality is demonstrated on a cardiac stress test (or equivalent local standard stress test). Participants with an abnormal cardiac stress test may be considered for study participation if they have adequate ejection fraction and cardiology clearance with approval of the Investigator.
* Patients who have obstructive or restrictive pulmonary disease and have a documented forced expiratory volume in 1 second (FEV1) of ≤ 60% of predicted normal:

  * If a patient is not able to perform reliable spirometry due to abnormal upper airway anatomy (i.e., tracheostomy), a 6-minute walk test may be used to assess pulmonary function.,
  * Patients who are unable to walk a distance of at least 80% predicted for age and sex or demonstrates evidence of hypoxia at any point during the test (SpO2 < 90%) are excluded.
* Patients who have had another primary malignancy within the previous three (3) years (with the exception of carcinoma in situ of the breast, cervix, or bladder; localized prostate cancer; non-melanoma skin cancer that has been adequately treated; or other cancers that in the opinion of the investigator do not place the subject at a significantly higher risk).
* Active infections, including COVID-19, within 30 days
* Participated in another clinical study with an investigational product within 21 days of the initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
LN-144 Efficacy | 1 year following TIL infusion
  measured as the rate of RFS (Relapse-Free Survival)
LN-144 Safety Profile | Within 30 days of LN-144 administration
  measured by the incidence Serous Adverse Events (SAE)

SECONDARY OUTCOMES:
LN-144+ Pembrolizumab Efficacy Overall Survival (OS) | 1 year after initial treatment
  measured using overall survival (OS). This is the length of time from the start of treatment to a given time point that measures participants on the study that are still alive
LN-144+ Pembrolizumab Efficacy Relapse-Free Survival (RFS) | 1 year after initial treatment
  measured using Relapse-free survival described as the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer
LN-144+ Pembrolizumab Efficacy Distant Metastasis-Free Survival (DMFS) | 1 year after inital treatment
  measured using distant metastasis-free survival (DMFS). This is the length of time from the start of treatment for cancer that a patient is still alive and the cancer has not spread to other parts of the body.
LN-144 Safety Profile | within 12 months of LN144 administration
  Incidence of adverse events following LN144 administration
Location of relapse | Up to 3 years
  In participants who relapse, the location of the relapse will be located using standard imaging and physical exam
Rate of Achievable Recruitment | 2 years from the study start date
  The number of participants enrolled will be counted in which an "achievable" recruitment is considered to be 1 participant every 2-3 months.

CONTACTS AND LOCATIONS:
Overall Officials: James Isaacs, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No